CLINICAL TRIAL: NCT02509468
Title: Treatment of Superficial Voluminous Complicated Slow-flow Vascular Malformations With Sirolimus: a Phase 2 Trial in Children Observational-phase Designed
Brief Title: suPERficial Slow-flow Vascular malFORMations Treated With sirolimUS
Acronym: PERFORMUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PHRN14-AM/PERFORMUS; 2015-001096-43 (EudraCT Number)
Record Dates: First submitted 2015-07-15; First posted 2015-07-28 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2019-09

CONDITIONS: Vascular Malformation
MeSH Terms: conditions — Vascular Malformations | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational (No Intervention): Patients will first be included in an observational period, then, at a randomized time different from one to another, will all receive the experimental treatment (i.e. sirolimus).
  This design has been defined a the "randomized placebo-phase design" (Feldman et al. J Clin Epidemiol. 2001 Jun;54(6):550-7)
- Experimental (Experimental): At a randomized date, patients will start treatment with sirolimus (beginning dose: 0.08mg/kg/day)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — * each patient will be followed during a 12-month-period
  * each patient will start by an observational period and end being treated by sirolimus
  * at a random date (between month 4 and month 8), each patient will switch from the observational period to the sirolimus period
  Other Names: rapamune
  Arms: Experimental

SUMMARY:
The most recent classification, adopted by International Society for the Study of Vascular Anomalies (ISSVA) in 1996, and updated in Melbourne in 2014, divides these lesions into two broad categories: vascular tumors and vascular malformations. Vascular malformations (VMs) are subdivided into high-flow VM and slow-flow VM.

Slow-flow VMs consist of congenital anomalies which may involve abnormal capillaries vessels, venous vessels, lymphatic vessels or combination of several of them. They can be superficial (involving cutaneous and subcutaneous tissues) and/or may have visceral involvement. They can be limited or diffuse, and are sometimes components of genetic hypertrophic syndromes.

The diagnosis of slow-flow VMs is performed on physical examination (biopsy may be required for confirmation), and is completed with imaging (ultrasonography and magnetic resonance imaging (MRI)). Slow-flow VMs may be particularly voluminous; associated with underlying hypertrophy responsible for functional impairment; painful; associated with seepage or continuous cutaneous bleeding; complicated with visceral signs or hematologic disturbances (anemia, thrombopenia). Management requires dedicated multispecialty care. There are no guidelines for treatment, and management may include no intervention - but natural history of these VMs is progressive worsening -, compression by physical bandage, sclerotherapy, resection (when feasible),anti-inflammatory or anti-coagulation drugs.

Case reports and series have provided evidence for supporting the need for a clinical trial of sirolimus by reporting successful treatment on several children with complicated vascular anomalies. The choice of sirolimus is rational. Mammalian target of rapamycin (mTOR) is a serine/threonine kinase regulated by phosphoinositide-3-kinase involved in cell mobility, cell growth and angiogenesis. Sirolimus inhibits mTOR, which induces inhibition of angiogenesis, in particular lymphangiogenesis, which has been demonstrated in several models.

DETAILED DESCRIPTION:
Vascular anomalies include a heterogeneous group of disorders of newborns and children. While infantile hemangioma are common (10% of infants), generally not complicated and easily managed, the majority of other vascular anomalies are rare (<2% altogether) and have no guidelines for management. The most recent classification, adopted by International Society for the Study of Vascular Anomalies (ISSVA) in 1996, divides these lesions into two broad categories: vascular tumors and vascular malformations. Vascular malformations (VMs) are subdivided into high-flow VM and slow-flow VM.

Slow-flow VMs consist of congenital anomalies which may involve abnormal capillaries vessels, venous vessels, lymphatic vessels or combination of several of them. They can be superficial (involving cutaneous and subcutaneous tissues) and/or may have visceral involvement. They can be limited or diffuse, and are sometimes components of genetic hypertrophic syndromes. They always result from defective embryologic vasculogenesis.

The diagnosis of slow-flow VMs is performed on physical examination - a biopsy may be required for confirmation -, and is completed with imaging, which includes ultrasonography and magnetic resonance imaging (MRI). Slow-flow VMs may be simple to manage or can be complicated for several reasons: they may be particularly voluminous; associated with underlying hypertrophy responsible for functional impairment; painful; associated with seepage or continuous cutaneous bleeding; complicated with visceral signs or hematologic disturbances (anemia, thrombopenia). Management requires dedicated multispecialty care. There are no guidelines for treatment, and management may include no intervention - but natural history of these VMs is progressive worsening -, compression by physical bandage, sclerotherapy, resection (when feasible), anti-inflammatory or anti-coagulation drugs.

The vast majority of literature reporting medical therapies consists of paediatric case reports, and is complicated by publication bias, inconsistent use of nomenclature and absence of clinical trials. Case reports and series have provided evidence for supporting the need for a clinical trial of sirolimus by reporting successful treatment on several children with complicated vascular anomalies. The choice of sirolimus is rational. Mammalian target of rapamycin (mTOR) is a serine/threonine kinase regulated by phosphoinositide-3-kinase involved in cell mobility, cell growth and angiogenesis. Sirolimus inhibits mTOR, which induces inhibition of angiogenesis, in particular lymphangiogenesis, which has been demonstrated in several models.

Randomized observational-phase design (Feldman et al. J Clin Epidemiol 2001;54:550-557):

* each patient will be followed during a 12-month-period
* each patient will start by an observational period and will end being treated by sirolimus
* at a random date (between month 4 and month 8), each patient will switch from the observational period to the sirolimus period Therefore, each patient will be his/her own control, as in a cross-over trial (but the difference is that the cross-over is all in one direction, from observational period to treatment period). This explains why variation in volume will be standardized by period durations.

As specified by Feldman et al, the randomized placebo-phase design is well adapted in situations where "a placebo controlled study would be perceived as being unacceptable by enrolling physicians and by patient" and "may be especially useful when highly potent therapies for rare diseases"

ELIGIBILITY:
* Patients aged from 6 years to 18 years
* With a slow-flow vascular malformation confirmed by MRI, included or not into a genetic disorder, among the following:
* microcystic lymphatic malformation
* mixed micro- and macrocystic malformation
* venous malformation
* combined lymphatic and venous malformation
* Malformation voluminous and complicated (pain, functional impairment, bleeding, seepage)
* Extended to the underlying subcutaneous tissue, to the fascias, the muscles and/or the underlying bone
* MRI of the VM performed within 8 months
* Vaccination schedule updated
* Informed, written consent of the subject's parents or the 18 years old subject
* Cooperative parent or subject, aware of the necessity and duration of controls so that perfect adhesion to the protocol could be expected
* Subjects or subject's parents covered by or having the rights to social security.

Exclusion criteria:

* Slow-flow VMs which are only macrocystic lymphatic malformations
* Visceral life-threatening involvement
* Patients who received prior per os treatment with an mTOR inhibitor
* Immunosuppression (immunosuppressive disease or immunosuppressive treatment)
* Known chronic infectious disease
* History of cancer in the 2 previous years
* Brest feeding or pregnant women, or women on childbearing age without effective contraception, up to 12 weeks after treatment discontinuation
* Known allergy to mTOR inhibitor
* Concomitant treatment that inhibits or activates CYP3A4, and P-gp glycoprotein, cytotoxic drugs, antilymphocyte immunoglobulines and metoclopramide
* Intolerance to fructose, intolerance or malabsorption to glucose, galactose, metabolic insufficiency in sucraseisomaltase, metabolic defect in lactase
* Known allergy to peanuts or soyabean
* Liver insufficiency (elevated transaminases > 2.5 N)
* Anemia with Hb < 9 g/dl
* Leukopenia < 1000/mm3
* Thrombocytopenia < 80 000/mm3
* Hypercholesterolemia (LDL-cholesterol ≥ 2g/l)
* Patients with risk of opportunistic infections
* Contraindication of MRI
* Known allergy to lidocaïne
* Live attenuated vaccine up to 3 months after sirolimus discontinuation
* Subject already participating to a therapeutic study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change of volume of the Vascular Malformation | at baseline, at date of switch from the observational period to the sirolimus period (between 4 and 8 month) and at 12 months
  Primary outcome will be based on the volume of the VMs on MRI. Three MRI will be performed: one at baseline (M0), one at the date of switch from the observational period to the sirolimus period (MS) and one at the end of follow-up (M12). Relative change of volume, standardized by the duration period, will define the outcome. Thus, for the observational period, the primary outcome is defined as {(VMS - V0)/V0}/(MS-M0) where V0 and VMS are the volumes assessed at baseline and month S, respectively, and (MS-M0) corresponds to the duration of the observational period. For the sirolimus period, the outcome is defined in the same way as {(V12 - VMS)/VMS}/(M12-MS), where V12 is the volume assessed at month 12 and (M12-MS) corresponds to the duration of the sirolimus period.
  Interpretation of the MRI will be centralized and performed by a radiologist blinded from physical assessment and from treatment period.

SECONDARY OUTCOMES:
Efficacy of study treatment measured on digital photographs | inclusion, switch from the observational period to the sirolimus period (between 4 and 8 month), switch+1month, 12 month
  Qualitative assessment of efficacy on digital photographs
Self assessment of efficacy of study treatment | Participants will be followed during 12 months
  Patient self assessment or proxy (parents) self assessments using visual analogic scale (0-10):
  * Global treatment efficacy on a visual analogic scale (0-10)
  * Skin complications/symptoms (seepage, bleeding, skin tension, functional impairment)
  * Pain
  * Quality of life by the dermatological quality of life scale (DLQI and DLQI adapted to children)
Dermatologist's assessment of efficacy of study treatment | Participants will be followed during 12 months
  Dermatologist's global assessment of efficacy using a visual analogic scale (0-10)
Efficacy of study treatment | Participants will be followed during 12 months
  Decrease of vascular endothelium growth factor (VEGF) and Tissue Factor (TF) plasma levels Platelet count, and fibrinogen, D-dimers, factor V levels supporting the presence and disappearance of an abnormal intravascular coagulation consumption
Adverse events and safe adverse events will be compared | Participants will be followed during 12 months
  Adverse events and safe adverse events will be compared using the Mc Nemar test, if applicable. Otherwise, descriptive statistics (percentages) will be estimated.
Organic collection of skin and blood samples | at 5 month or 6 month or 7 month or 8 month or 9 month after inclusion
  From the organic collection (including blood and skin samples), genetic analysis of several genes involved in vasculogenesis (currently TIE2 and PIK3CA) will be performed. A genotype/phenotype study will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Maruani, MD, PhD, Principal Investigator — CHRU TOURS
Locations (12):
- France (12):
  - Service de dermatologie, CHU Angers, Angers
  - Service de dermatologie, Hôpital du Bocage, CHU Dijon, Dijon
  - Explorations Médecine Vasculaire Hôpital A. Michallon, CHU de Grenoble, Grenoble
  - Service de radiologie Hôpital Femme-Mère-Enfant, Hospices Civils de Lyon, Lyon
  - Service de Dermatologie, vénéréologie et cancérologie cutanée, Hôpital La Timone APHM, Marseille
  - Service de Dermatologie, Hôpital St Eloi, CHU Montpellier, Montpellier
  - Service de Dermatologie, Hôpital Hôtel-Dieu, CHU Nantes, Nantes
  - Service de dermatologie, CHU Nice, Nice
  - Service de dermatologie, APHP Necker, Paris
  - Service de Dermatologie, Hôpital Pontchaillou, CHU RENNES, Rennes
  - Service de dermatologie, Hôpital Larrey, CHU Toulouse, Toulouse
  - Consultations externes de Dermatologie, Hôpital Clocheville, CHU Tours, Tours

REFERENCES:
- [Result] Maruani A, Tavernier E, Boccara O, Mazereeuw-Hautier J, Leducq S, Bessis D, Guibaud L, Vabres P, Carmignac V, Mallet S, Barbarot S, Chiaverini C, Droitcourt C, Bursztejn AC, Lengelle C, Woillard JB, Herbreteau D, Le Touze A, Joly A, Leaute-Labreze C, Powell J, Bourgoin H, Gissot V, Giraudeau B, Morel B. Sirolimus (Rapamycin) for Slow-Flow Malformations in Children: The Observational-Phase Randomized Clinical PERFORMUS Trial. JAMA Dermatol. 2021 Nov 1;157(11):1289-1298. doi: 10.1001/jamadermatol.2021.3459. PMID 34524406
- [Derived] Maruani A, Boccara O, Bessis D, Guibaud L, Vabres P, Mazereeuw-Hautier J, Barbarot S, Chiaverini C, Blaise S, Droitcourt C, Mallet S, Martin L, Lorette G, Woillard JB, Jonville-Bera AP, Rollin J, Gruel Y, Herbreteau D, Goga D, le Touze A, Leducq S, Gissot V, Morel B, Tavernier E, Giraudeau B; Groupe de Recherche de la Societe Francaise de Dermatologie Pediatrique. Treatment of voluminous and complicated superficial slow-flow vascular malformations with sirolimus (PERFORMUS): protocol for a multicenter phase 2 trial with a randomized observational-phase design. Trials. 2018 Jun 27;19(1):340. doi: 10.1186/s13063-018-2725-1. PMID 29945674